CLINICAL TRIAL: NCT00538369
Title: Combining Observational and Physiologic Sedation Assessment Tools
Acronym: COST
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of equipoise
Sponsor: Duke University (Other)
Collaborators: University of North Carolina (Other); Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00008519; 8771-06 - 8RO
Record Dates: First submitted 2007-10-01; First posted 2007-10-02 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2007-10

CONDITIONS: Brain Injury
Keywords: Nursing; critical care; sedation assessment; Bispectral index
MeSH Terms: conditions — Brain Injuries | interventions — Consciousness Monitors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard-of-care (Active Comparator): The standard-of-care group will receive sedation assessment and monitoring with the Ramsay scale, which is the accepted tool at this university
  Interventions: Other: Ramsay Scale
- standard + BIS (Experimental): Subjects in the standard-of-care + BIS group will receive sedation assessment and monitoring using the Ramsay scale and values from the bispectral index (BIS) monitor.
  Interventions: Other: Ramsay Scale; Device: Bispectral index monitor

INTERVENTIONS:
Other: Ramsay Scale — While receiving sedation, subjects will be monitored with the Ramsay scale
  Other Names: Ramsay sedation scale
Device: Bispectral index monitor — While receiving sedation, subjects will receive BIS monitoring
  Other Names: BIS
  Arms: standard + BIS

SUMMARY:
When a physiologic tool to measure the patient's hypnotic state is added to current practice tools is there a decrease in the amount of drug the patient receives.

DETAILED DESCRIPTION:
The purposes of this study were to examine the effect of combining a physiologic measure of consciousness (BIS) with observational assessment of sedation (Ramsay) on infused sedation drug volumes, undersedation events, and the recovery time to arouse from sedation, in a group of neurocritically ill patients. During a 12-hour data collection period, patients received sedation assessment and management with either the current standard of care (sedation assessment with the Ramsay scale), or the standard of care plus the addition of physiologic data from BIS monitoring. Planned research questions explored how BIS monitoring impacts short-term sedation-related outcomes.

Research Questions

* Is there less sedation drug use for patients when nurses monitor sedation with BIS augmentation of Ramsay than when nurses monitor patients with Ramsay alone?
* Is sedation assessment augmented by BIS use associated with a decreased time to wake-up (recovery time) when nurses are instructed to interrupt sedation and obtain a neurologic examination, compared to use of Ramsay alone?
* Are there differences in the number of events associated with undersedation (e.g., self-extubation) for patients assigned to BIS augmentation compared to patients assigned to Ramsay alone?

ELIGIBILITY:
Inclusion Criteria:

* Adult
* admitted with a neurological or neurosurgical diagnosis
* intubated and on mechanical ventilatory support
* receiving continuous sedation with propofol
* Glasgow Coma Score <12

Exclusion Criteria:

* bifrontal brain injury
* status epilepticus
* barbiturate coma therapy
* continuous benzodiazepine administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2006-11; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
How much sedative was infused | length of stay

SECONDARY OUTCOMES:
How quickly the subject recovered from sedation | once
The number of undersedation events | length of stay in ICU

CONTACTS AND LOCATIONS:
Overall Officials: DaiWai M Olson, PhD RN CCRN, Principal Investigator — Duke University; Suzanne M Thoyre, PhD RN, Study Chair — University of North Carolina, Chapel Hill; Carmelo Graffagnino, MD FRCPC, Study Director — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Ramsay MA, Savege TM, Simpson BR, Goodwin R. Controlled sedation with alphaxalone-alphadolone. Br Med J. 1974 Jun 22;2(5920):656-9. doi: 10.1136/bmj.2.5920.656. PMID 4835444